CLINICAL TRIAL: NCT05896488
Title: A Study to Assess the Sweat Response, Sweat Composition and Thermoregulatory Response to Exercise in Heat in Adults With Cystic Fibrosis on Cystic Fibrosis Transmembrane Conductance Regulator Modulator Therapy Compared Healthy Controls.
Brief Title: Sweat Response, Sweat Composition and Thermoregulatory Response to Exercise in Heat in Adults With Cystic Fibrosis on Modulator Therapy.
Acronym: Sweat-CF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Portsmouth (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Reader (Associate Professor) in Clinical Exercise Physiology, University of Portsmouth
Other Study IDs: 315193
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Cystic Fibrosis
Keywords: Exercise, CFTR modulator therapy, thermoregulation, heat-related illness, sweat sodium
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis: No intervention - only assessments
- Healthy Control: No intervention- only assessments

SUMMARY:
Cystic fibrosis (CF) is a common inherited condition in the Caucasian population resulting in poor function and/or production of the CF transmembrane conductance regulator (CFTR) protein. The CFTR protein plays a crucial role in the secretion and re-absorption of sodium chloride within the sweat gland. The sweat gland has played a key role in diagnosing and understanding CF with sweat chloride elevation being a key criterion to diagnosing CF. People with CF are thought to be at risk of exertional heat illness during exposure to hot environments or during prolonged periods of exercise and are currently encouraged to take salt supplements during periods of excessive sweating.

Kaftrio®, a newly approved pharmacological therapy has shown a rapid and sustained reduction in sweat chloride levels on initiation of this treatment. This study will aim to play a crucial part in understanding the sweat response, sweat composition and the thermoregulatory response to exercise in the heat in people with CF on Kaftrio®.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a common inherited condition in the Caucasian population, affecting approximately 52, 246 people in Europe. Mutations in the CF transmembrane conductance regulator (CFTR) gene results in poor function or production of the CFTR protein which functions as an anion channel to transport ions across the cell membrane.

The sweat gland has played a substantial part in diagnosing and understanding CF with sweat chloride elevation being a key criterion to diagnosing CF. Traditionally, abnormal function of the CFTR protein in the sweat gland results in failure to reabsorb sodium chloride leading to excessive salt loss. People with CF are thought to be at risk of exertional heat illness during exposure to hot environments or during prolonged periods of exercise and are currently encouraged to take salt supplements during periods of excessive sweating.

Over the last decade pharmacological therapies (CFTR modulator therapies (CFTRm)) which target the underlying cellular defect characterising CFTR in people with CF have been developed. Kaftrio® is now the most widely used modulator therapy. Studies have shown a rapid and sustained reduction in sweat chloride levels on initiation of these highly effective CFTRm. The need for salt supplementation may be influenced when taking CFTRm. Therefore, there is a need to further understand the sweat response relative to the needs in people with CF.

This study will recruit 9 people with CF who currently taking Kaftrio® and 9 healthy age-, sex- and weight-matched controls who are ≥ 18 years old. We will ask all participants to attend the laboratories for 2 visits. Visit 1 is designed to calculate metabolic heat production during different cycling intensities in order to set the workload for visit 2 relative to their metabolic heat production. Visit 2 is designed to collect sweat and thermoregulatory indices during 1 hour of cycling in the heat.

This study will compare the sweating and thermoregulatory response to exercising in the heat in a group of people with CF who are stable on Kaftrio® compared to a healthy matched control group.

The aims of this study are to:

1. Determine the sweat sodium concentration in adults with CF on Kaftrio® from exercise at a fixed-rate of metabolic heat production under heat stress conditions and whether this is different to healthy age- weight- and sex- matched controls;
2. Determine the local and whole-body sweat rate in adults with CF on Kaftrio® during exercise under heat stress conditions and whether this is different to healthy age- weight- and sex- matched controls;
3. Determine how adults with CF on Kaftrio® respond in terms of skin blood flow during exercise under heat stress conditions and whether this is different to healthy age- weight- and sex- matched controls;
4. Determine thermal strain from skin and core body temperature in adults with CF on Kaftrio® during exercise under heat stress conditions and whether this is different to healthy age- weight- and sex- matched controls.

ELIGIBILITY:
Inclusion Criteria for participants with CF:

* Is taking CFTRm
* Males and females ≥ 18 years of age
* CF diagnosis based on clinical features, supported by a history of an abnormal sweat test (sweat [Cl-] > 60 mmol·L-1 > 100 mg sweat), where possible, diagnostic genotyping would also be desired
* Can clearly state that they are not pregnant
* No contraindications to performing exhaustive exercise
* Can understand and cooperate with the study protocol
* No exacerbation (increase in cough, sputum or breathlessness, or change in the colour of sputum) within the preceding 2 weeks
* No weight loss in the preceding 2 weeks

Inclusion Criteria for healthy control participants:

* Healthy males and females who are age- weight- and sex- matched to the enrolled individuals with CF
* Can clearly state that they are not pregnant
* No clinical diagnosis of a chronic disease
* Can understand and cooperate with the study protocol
* No contraindications to performing exhaustive exercise

Exclusion Criteria for participants with CF:

* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders (arthritis, joint or muscle disease) and cardiovascular disease (congenital heart disease or cardiomyopathy).
* Unstable co-morbid asthma (daily pulmonary function variability of >20%)
* Is pregnant during the initial screening process
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not of a suitable age for testing
* Is a smoker or inhales any other substances

Exclusion Criteria for healthy control participants:

* Any pulmonary, metabolic or cardiovascular conditions
* Any other diagnosed disease
* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders (active arthritis, joint or muscle disease) and cardiovascular disease (congenital heart disease or cardiomyopathy)
* Is pregnant during the initial screening process
* Presents with co-morbidities to performing exhaustive exercise
* Is a smoker or inhales any other substances
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not an age- weight- or sex-match for the CF group

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from adult CF outpatient clinics within the CF network. If a potential participant outside of the CF network wishes to participant they will be screened by the CF consultants within the CF network.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2023-03-18 (Actual); Primary Completion 2024-03-18 (Estimated); Study Completion 2024-03-18 (Estimated)

PRIMARY OUTCOMES:
Sweat sodium concentration (mmol∙L-1) | Day 2 - baseline
  Between group differences in sweat sodium concentration

SECONDARY OUTCOMES:
Whole-body sweat rate (mL) | Day 2 - baseline
  Between group differences in whole-body sweat rate derived from pre - post nude body mass
Forearm sweat rate (mg∙min-1∙cm2) | Day 2 - baseline
  Between group differences in forearm sweat rate
Mid-back sweat rate (mg∙min-1∙cm2) | Day 2 - baseline
  Between group differences in mid-back sweat rate
Sweat gland activity (gland∙cm2) | Day 2 - baseline
  Between group differences in sweat-gland activation derived from the modified-iodine patch technique
Core temperature (°C) | Day 2 - baseline
  Between group differences in core temperature derived from rectal temperature
Mean skin temperature (°C) | Day 2 - baseline
  Between group differences in skin temperature
Heart rate (b∙min-1) | Day 2 - baseline
  Between group differences in heart rate
Cutaneous blood flux | Day 2 - baseline
  Between group differences in cutaneous blood flux
Urine osmolality (mOsmol/kg) | Day 2 - baseline
  Between group differences in urine osmolality
Perception of temperature sensation | Day 2 - baseline
  Between group differences in perception of temperature sensation
Perception of thermal comfort | Day 2 - baseline
  Between group differences in perception of thermal comfort
Change in thermal comfort | Day 2 - baseline
  Between group differences in change in thermal comfort
Rate of change in thermal comfort | Day 2 - baseline
  Between group differences in rate of change in thermal comfort
Heat sensitivity | Day 2 - baseline
  Between group differences in heat sensitivity derived from sweat rate / change in thermal comfort
Heat illness symptom index | Day 2 - baseline
  Between group differences in heat-related illness symptoms
Maximal oxygen uptake (VO2 max) | Day 1 - baseline
  Between group differences in oxygen uptake derived from a maximal cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Portsmouth, Portsmouth, United Kingdom